CLINICAL TRIAL: NCT02409160
Title: Sleep, Pulmonary Function, Systemic and Adipose Immune Response and Quality of Life in Severe Obese Patients Undergoing Bariatric Surgery. A Protocol of Randomized Controlled Clinical Trial
Brief Title: Sleep and Immune Response in Severe Obese Patients Undergoing Bariatric Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário de Anapolis (Other)
Collaborators: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other); Clínica de Gastroenterologia e Medicina Avançada - GASTROMED (Unknown); Santa Casa de Misericórdia de Anápolis (Unknown)
Responsible Party: Principal Investigator, Luis Vicente Franco de Oliveira, Professor, Centro Universitário de Anapolis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 220506/2009
Record Dates: First submitted 2015-03-24; First posted 2015-04-06 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Severe Obesity; Morbid Obesity
Keywords: Severe Obesity; Sleep Disorders; Bariatric Surgery; Inflammation; Quality of Life
MeSH Terms: conditions — Obesity, Morbid; Sleep Wake Disorders; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bariatric Surgery (Experimental): Standard laparoscopic Roux-en-Y gastric bypass technique resulting in a gastric pouch with a volume of about 25 mL, a 100-cm-long Roux-limb, and a 75-cm-long biliopancreatic limb.
  Interventions: Procedure: Standard Roux-en-Y gastric bypass
- Control Group (No Intervention)

INTERVENTIONS:
Procedure: Standard Roux-en-Y gastric bypass
  Arms: Bariatric Surgery

SUMMARY:
Obesity is a major public health problem in developed and developing countries, causing a range of respiratory and metabolic changes. There is a strong correlation between obesity and cardiorespiratory sleep disorders. The weight loss reduces the comorbidities and improves the quality of life, but clinical treatment it is not effective for a long period. In this context, currently bariatric surgery is an option for the real weight loss in the long term. Obstructive sleep apnea (OSA) is a common clinical condition observed in patients with obesity. The primary aim of this protocol are to assess the inflammatory profile of severe obese patients undergone to bariatric surgery, through systemic and adipose markers of inflammation. A secondary objective is study the impact of this surgery on sleep variables and quality of life. Investigators hypothesized that weight loss induced by bariatric surgery reduces systemic inflammatory profile, improve sleep quality and quality of life of subjects with severe obesity. Will participate in this study, patients with severe obesity (BMI > 40 or 35 to 39.9 kg/m2 associated comorbidities), with indication of bariatric surgery, screened Bariatric Surgery Service of Santa Casa de São Paulo in São Paulo. Inclusion criteria are severely obese, bariatric surgery indication and agreement to participate in the study. Are excluded patients with BMI > 55 kg/m2, clinical instability, mental instability or significant and unrealistic expectations of surgery. Patients will be assessed before and after bariatric surgery, 90, 180 and 360 days. The evaluation protocol will consist of clinical history, vital signs, neck and waist circumference, clinical analysis of blood inflammatory markers, lung function tests, maximal ventilatory pressures, full overnight standard polysomnography, excessive daytime sleepiness scale, cardiovascular risk, quality of life and personal satisfaction questionnaires.

DETAILED DESCRIPTION:
Obesity is a major public health problem in developed and developing countries, causing a range of respiratory and metabolic changes. There is a strong correlation between obesity and cardiorespiratory sleep disorders. The weight loss reduces the comorbidities and improves the quality of life, but clinical treatment it is not effective for a long period. In this context, currently bariatric surgery is an option for the real weight loss in the long term. Obstructive sleep apnea (OSA) is a common clinical condition observed in patients with obesity. Recent studies have found that more than 2/3 of obese patients also have OSA, and that these exhibit similar pathophysiological substrates for cardiovascular disease where increased blood pressure is a common consequence. This raises another discussion where obesity and OSA may have an additive effect on cardiovascular risk factors. Our main objective is to evaluate whether the systemic and adipose markers of inflammation alters after bariatric surgery through biochemical indexes in the visceral (omental, mesenteric) and subcutaneous adipose tissue depots and fasting blood samples, including the proinflammatory cytokines tumor necrosis factor α (TNFα), interleukin 6 (IL-6), interleukin 8 (IL-8), interleukin 18 (IL-18), soluble TNF receptor-2 (sTNFR2), soluble E-selectin, soluble intercellular adhesion molecule-1 (sICAM-1), soluble vascular cell adhesion molecule-1 (sVCAM-1), monocyte chemoattractant protein 1 (MCP 1), high sensitivity C-reactive protein (hsCRP), adiponectin (AdipoQ) genes, vascular endothelial growth factor A (VEGF-A), nuclear factor Kappa B (NF-kB) and adipose-derived hormone leptin. Moreover, identify the possible association of systemic and adipose inflammation before bariatric surgery with the magnitude of surgery-induced weight loss and to assess pulmonary function through spirometry and, maximal ventilatory pressures through vacuometry; to determine whether surgical procedure induced decrease in body weight, BMI, abdominal circumference and, improve quality of life; to study sleep patterns through full standard polysomnography and quality of life in obese patients undergone to bariatric surgery and verify a possible correlation between weight loss and physiological variables. Will participate in this study, patients with severe obesity (BMI > 40 or 35 to 39.9 kg/m2 associated comorbidities), with indication of bariatric surgery, screened Bariatric Surgery Service of Santa Casa de São Paulo in São Paulo. Inclusion criteria are severely obese, bariatric surgery indication and agreement to participate in the study. Are excluded patients with BMI > 55 kg/m2, clinical instability, mental instability or significant and unrealistic expectations of surgery. Patients will be assessed before and after bariatric surgery, 90, 180 and 360 days. The evaluation protocol will consist of clinical history, vital signs, neck and waist circumference, clinical analysis of blood inflammatory markers, lung function tests, maximal ventilatory pressures, full overnight standard polysomnography, excessive daytime sleepiness scale, cardiovascular risk, quality of life and personal satisfaction questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients eligible for the trial must comply with all of the following at randomization:
2. male and female patients aged 18 to 65 years,
3. grade III severe obesity (BMI ≥ 40 kg/m2) or ≥ 35 kg/m2 with comorbidities,
4. awaiting bariatric surgery,
5. with documented history of conventional weight loss attempts having proven unsuccessful over time,
6. and if they are able to understand and agreement to participate in the study through a signed term of informed consent.

Exclusion Criteria:

1. Any medical condition rendering surgery too risky;
2. BMI above 55 kg/m2;
3. Unrealistic postoperative target weight and/or unrealistic expectations of surgical treatment;
4. Pregnancy, lactation or planned pregnancy within two years of potential surgical treatment;
5. Lack of safe access to abdominal cavity or gastrointestinal tract;
6. Abusive alcohol use or drug use.
7. Cancer
8. Any cardiorespiratory condition opposite indicate the surgical procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in systemic immune response after bariatric surgery. | Baseline immune response to 180 days.
  Systemic markers of inflammation through fasting blood samples biochemical indexes.
Change in systemic adipose inflammation response after bariatric surgery. | Baseline adipose inflammation response to 180 days.
  Systemic markers of inflammation through biochemical indexes in the visceral (omental, mesenteric) and subcutaneous adipose tissue depots.

SECONDARY OUTCOMES:
Alterations in sleep quality after bariatric surgery. | 180 days
  Study sleep patterns through full standard polysomnography.
Changes in pulmonary function after bariatric surgery. | 180 days
  Assess pulmonary function through spirometry.
Changes in maximal ventilatory pressures after bariatric surgery. | 180 days
  Assess maximal inspiratory and expiratory pressures through vacuometry.
Changes in health related quality of life after bariatric surgery. | 180 days
  Changes in quality of life through Short Form-36 and BAROS questionnaires.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Gastromed, Anápolis, Goiás
  - Centro Universitário de Anápolis - UniEVANGÉLICA, Anápolis, Goiás
  - Department of Surgery of Santa Casa of São Paulo Medical School, Gastric Surgery Division, São Paulo, São Paulo

REFERENCES:
- [Derived] Felipe LA, Bachi ALL, Oliveira MC, Moreira SMBP, Afonso JPR, Lino MEM, Paixao V, Silva CHM, Vieira RP, Vencio S, Jirjos EI, Malheiros CA, Insalaco G, Junior WRF, Oliveira LVF. Effects of Roux-en-Y gastric bypass on the metabolic profile and systemic inflammatory status of women with metabolic syndrome: randomized controlled clinical trial. Diabetol Metab Syndr. 2023 Feb 14;15(1):19. doi: 10.1186/s13098-023-00986-2. PMID 36788619
- [Derived] de Sousa ART, Freitas Junior WR, Perez EA, Ilias EJ, Silva AS, Alves VLS, Afonso JPR, Oliveira MC, Fonseca AL, da Silva MM, Lino MEM, Oliveira Junior MC, Vieira RP, Pedro WJS, Bachi ALL, Insalaco G, Malheiros CA, Oliveira LVF. Surgery for Obesity and Weight-Related Diseases Changes the Inflammatory Profile in Women with Severe Obesity: a Randomized Controlled Clinical Trial. Obes Surg. 2021 Dec;31(12):5224-5236. doi: 10.1007/s11695-021-05702-5. Epub 2021 Sep 23. PMID 34554379
- [Derived] Perez EA, Oliveira LVF, Freitas WR Jr, Malheiros CA, Ilias EJ, Silva AS, Urbano JJ, Oliveira PC, Cepeda FX, Sampaio LMM, Trombetta IC, Delle H, Neto DG, Nacif SR, Stirbulov R. Prevalence and severity of syndrome Z in women with metabolic syndrome on waiting list for bariatric surgery: a cross-sectional study. Diabetol Metab Syndr. 2017 Sep 20;9:72. doi: 10.1186/s13098-017-0269-2. eCollection 2017. PMID 28943894